CLINICAL TRIAL: NCT00306215
Title: A Multinational, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of CCX282-B in Subjects With Moderate to Severe Crohn's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of CCX282-B in Subjects With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL004_282
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Crohn's Disease
Keywords: double-blind; placebo-controlled; multicenter; efficacy; safety
MeSH Terms: conditions — Crohn Disease | interventions — CCX282-B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Blinded study arm
  Interventions: Drug: CCX282-B
- 2 (Experimental): Blinded study arm
  Interventions: Drug: CCX282-B
- 3 (Experimental): Blinded study arm
  Interventions: Drug: CCX282-B
- 4 (Experimental): Blinded study arm
  Interventions: Drug: CCX282-B

INTERVENTIONS:
Drug: CCX282-B — CCX282-B or placebo capsules

SUMMARY:
The purpose of this study is to determine whether CCX282-B is effective in treating patients with moderate to severe Crohn's Disease.

DETAILED DESCRIPTION:
Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Key Inclusion Criteria:

* moderate to severe Crohn's Disease
* CDAI 250-450
* CRP >7.5
* signed written informed consent

Key Exclusion Criteria:

* > 100 cm of small bowel resected
* ileostomy, colostomy or rectal pouch
* diagnosis of ulcerative colitis or indeterminate colitis
* evidence of short bowel syndrome requiring enteral or parenteral supplementation or total parenteral nutrition
* hepatitis B, C or HIV infection
* history of infection requiring IV antibiotics
* serious or GI infection in the previous 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving a clinical response (defined as a decrease from baseline in Crohn's Disease Activity Index [CDAI] score of at least 70) on Day 57 | Day 57

SECONDARY OUTCOMES:
Percentage of subjects achieving clinical remission (defined as a Crohn's Disease Activity Index [CDAI] score less than or equal to 150) on Day 57 | Day 57

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (112):
- Australia (11):
  - Bankstown - Lidcombe Hospital, Bankstown, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincents Hospital, Fitzroy, Victoria
  - Bayside Gastroenterology, Frankston, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Alfred Hospital, Prahran, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Austria (5):
  - Universitätsklinik für Innere Medizin, Innsbruck
  - A.ö. Krankenhaus der Elisabethinen Linz, Linz
  - Landesklinikum St. Poelten, Pölten
  - Krankenanstalt Rudolfstiftung, Vienna
  - Universitätsklinik für Innere Medizin III, Vienna
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
- Brazil (13):
  - Unigastro, Campinas
  - Centro Petropolitano de Reumatologia e Fisioterapia, Centro Petrópolis
  - Hospital das Clínicas de Curitiba UFPR, Curitiba
  - Hospital Geral de Goiânia, Goiânia
  - Instituto Goiano de Gastro, Goiânia
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital São Lucas PUC-RS, Porto Alegre
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro
  - Santo André Diagnósticos e tratamentoLtda., Santo André
  - Irmandade da Santa Casa de Misericórdia de Santos, Santos
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo
  - Hospital das Clínicas de São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
- Bulgaria (7):
  - 4 MHAT, 38 "Makedonia" 1000, Sofia
  - Military Medical Academy, Sofia
  - UMHAT "Alexandrovska", Sofia
  - UMHAT Queen Joanna, Sofia
  - UMHAT" St. Ivan Rilsky", Sofia
  - V City Hospital, Sofia
  - UMHAT "St. Marina", Varna
- Canada (8):
  - Health Science Centre, Calgary, Alberta
  - Lair Centre, Vancouver, British Columbia
  - DHC Research, Richmond Hill, Ontario
  - Mt. Sinai Hospital, Toronto, Ontario
  - Centre Hospitalier--Hotel-Dieu de Levis, Lévis, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHAUQ-Hopital St-Sacrement, Québec, Quebec
- Czechia (9):
  - Private Gastroenterology Centre, České Budejovice
  - Hepato-Gastroenterologie, Edvarda Benese 1549, Hradec Králové
  - II.Interni klinika, Endoskopie, Olomouc
  - Fakultni nemocnice, Prague
  - Klinika hepatogastroenterologieIKEM, Prague
  - General University Hospital Prague, Prague
  - Medic Kral ltd., Prague
  - Regional Hospital Pribram, Příbram
  - Regional Hospital Tabor, Tábor
- Denmark (4):
  - Medical Department V Århus University Hospital, Arhus C
  - Herlev Hospital Gastroenterologisk department, Herlev
  - Hvidovre Hospital, Hvidovre
  - Medical department S Odense University hospital, Odense
- France (5):
  - CHU Amiens - Hôpital Nord, Amiens
  - Service d'Hépato-Gastroentérologie et de Nutrition Clinique, Nice
  - Hopital du Haut-Lévêque, Pessac
  - Hôpital Charles Nicolle, Rouen
  - Service de Gastro-Enterologie et Nutrition, Toulouse
- Germany (7):
  - Charité Campus Mitte, Universitätsmedizin Berlin, Berlin
  - Medizinische Klinik m.S. Hepatologie, Gastroenterologie, Endokrinologie und Stoffwechsel, Berlin
  - Fachärztin für Innere Medizin, Hamburg
  - Klinikum der Christian-Albrechts-Universität zu Kiel, Kiel
  - Universitätsklinikum Magdeburg A.ö.R, Magdeburg
  - Gastroenterologische Praxis am Germania-Campus, Münster
  - Klinikum der Universität Regensburg, Regensburg
- Hungary (6):
  - Réthy Pál Kórház, Békéscsaba
  - Fővárosi Önkormányzat Bajcsy-Zsilinszky Kórház, Budapest
  - Debreceni Egyetem OEC, Debrecen
  - Vaszary Kolos Kórház, Esztergom
  - Petz Aladár Megyei Oktató Kórház, Győr
  - BAZ Megyei Kórház, Miskolc
- Israel (9):
  - Soroka Medical Center, Beersheba
  - Bnai Zion MC, Haifa
  - Rambam Medical Center,, Haifa
  - Hadassah Ein-Karem Medical Center, Jerusalem
  - Meir Hospital, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - The Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Trzifin
- Netherlands (3):
  - Ringweg Randenbroek 110, Amersfoort
  - Ikazia Ziekenhuis, Rotterdam
  - Isala Klinieken Locatie Sophia Afd. Interne Geneeskunde, Zwolle
- Poland (12):
  - ZOZ MSWiA Oddział Chorób Wewnętrznych, Bialystok
  - 10 Wojskowy Szpital Klinicznym, Oddzial Kliniczny Gasteroenterologii, Bydgoszcz
  - SPZOZ Wojewodzki Szpital, Bydgoszcz
  - Klinika Chorob Wewnetrznych I Gastroenterologii, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 4, Lublin
  - SPZOZ Szpital Wojewódzki w Opolu, Opole
  - SOPMED Niepubliczny Zakład Opieki Zdrowotnej, Sopot
  - Klinika Gastroenterologii i Chorób Wewnętrznych Samodzielny Publiczny Szpital Kliniczny nr 1 im. T. Sokołowskiego Pomorskiej Akademii Medycznej ul.Unii Lubelskiej 1, Szczecin
  - NZOZ Vivamed Zespół Lekarzy Specjalistów ul. Trocka 10A, Warsaw
  - CSK MSWiA, Klinika Gastroenterologii, Warsaw
  - Wojskowy Insytutu Medyczny, Warsaw
  - Klinika Gastroenterologii i Hepatologii, Akademii Medycznej, Wroclaw
- South Africa (5):
  - Panorama Medi Clinic, Cape Town
  - Louis Leipoldt Gastroenterology Centre, Louis Leipoldt Medical Centre, Cape Town
  - GastroEnterology Unit, Groote Schuur Hospital, Cape Town
  - Quatro Clinical Trial Institute, Cape Town
  - 427 Ontdekkers Road, Florida Park, Johannesburg
- Sweden (4):
  - Medicinkliniken, SU/Östra sjukhuset, Gothenburg
  - Universitetssjukhuset, Lund
  - Medicinmottagningen, Södersjukhuset, Stockholm
  - Sophiahemmet, Stockholm
- United Kingdom (2):
  - Centre for Gastroenterology Royal Free Hospital, London
  - Dept of Gastroenterology, John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Keshav S, Vanasek T, Niv Y, Petryka R, Howaldt S, Bafutto M, Racz I, Hetzel D, Nielsen OH, Vermeire S, Reinisch W, Karlen P, Schreiber S, Schall TJ, Bekker P; Prospective Randomized Oral-Therapy Evaluation in Crohn's Disease Trial-1 PROTECT-1 Study Group. A randomized controlled trial of the efficacy and safety of CCX282-B, an orally-administered blocker of chemokine receptor CCR9, for patients with Crohn's disease. PLoS One. 2013;8(3):e60094. doi: 10.1371/journal.pone.0060094. Epub 2013 Mar 20. PMID 23527300